CLINICAL TRIAL: NCT05396092
Title: The Effects of an Integrated Mindfulness-based Tai Chi Chuan Program on Sleep Disturbance Among Community-dwelling Elderly People: A Randomized Controlled Trial
Brief Title: The Effects of an Integrated Mindfulness-based Tai Chi Chuan Program on Sleep Disturbance Among Community-dwelling Elderly People
Acronym: MBTCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20210331002-01
Record Dates: First submitted 2022-05-17; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Elderly; Sleep; Mindfulness; Tai Chi Chuan
MeSH Terms: interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Integrated mindfulness-based Tai Chi Chuan (Experimental): MBTCC
  Interventions: Behavioral: Integrated mindfulness-based Tai Chi Chuan
- Mindfulness-based intervention (Active Comparator): MBI
  Interventions: Behavioral: Mindfulness-based intervention
- Tai Chi Chuan (Active Comparator): TCC
  Interventions: Behavioral: Tai Chi Chuan
- Sleep Hygiene Education (Active Comparator): SHE
  Interventions: Behavioral: Sleep Hygiene Education

INTERVENTIONS:
Behavioral: Integrated mindfulness-based Tai Chi Chuan — MBTCC will integrate components from both the MBI and TCC groups. The entire intervention consists of eight weekly sessions of two-and-a-half to three hours each.
  Other Names: MBTCC
  Arms: Integrated mindfulness-based Tai Chi Chuan
Behavioral: Mindfulness-based intervention — The MBI group is mainly based on the basic theory and research of the foundational mindfulness-based stress reduction program. The intervention consists of eight weekly sessions of two to two-and-a-half hours each.
  Other Names: MBI
  Arms: Mindfulness-based intervention
Behavioral: Tai Chi Chuan — TCC is mainly based on a nine-form Yang-style form of TCC, which is a brief and modified version of 64-form Yang-style TCC. The entire intervention consists of eight weekly sessions of two to two-and-a-half hours each.
  Other Names: TCC
  Arms: Tai Chi Chuan
Behavioral: Sleep Hygiene Education — SHE is based on principles used in stimulus control and sleep hygiene education, which has previously been used as the control group in sleep-related research. The entire intervention consists of eight weekly sessions of two to two-and-a-half hours each.
  Other Names: SHE
  Arms: Sleep Hygiene Education

SUMMARY:
The trial aims to evaluate the effects of an integrated form of mindfulness-based Tai Chi Chuan (MBTCC) program and the underlying mechanisms of the beneficial effects on sleep disturbance over 12-month follow-up in community-dwelling elderly people.

ELIGIBILITY:
Inclusion criteria:

* Aged 60 years or above;
* Classified as experiencing sleep disturbances (indication of poor sleep quality through a score >5 in the Pittsburgh Sleep Quality Index);
* Primary education level or above and able to communicate in Cantonese;
* Able to give informed consent; and
* No previous experience with meditation or other mind-body techniques (e.g., tai chi or yoga).

Exclusion criteria:

• Comorbid diagnoses of schizophrenia, schizoaffective disorder, substance misuse, organic brain syndrome, or intellectual disabilities.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-04-18 (Estimated); Study Completion 2025-04-18 (Estimated)

PRIMARY OUTCOMES:
the Insomnia Severity Index | at baseline (T1)
  This is a seven-item self-report questionnaire. A higher score represents greater insomnia severity.
the Insomnia Severity Index | In the 8th week from baseline (T2)
  This is a seven-item self-report questionnaire. A higher score represents greater insomnia severity.
the Insomnia Severity Index | six months after T2 (T3)
  This is a seven-item self-report questionnaire. A higher score represents greater insomnia severity.
the Insomnia Severity Index | one year after T2 (T4)
  This is a seven-item self-report questionnaire. A higher score represents greater insomnia severity.

SECONDARY OUTCOMES:
the Multidimensional Assessment of Interoceptive Awareness scale | at baseline (T1)
  The scale consists of 32 items and comprises eight subscales. A higher score indicates higher levels of interoceptive awareness.
the Multidimensional Assessment of Interoceptive Awareness scale | In the 8th week from baseline (T2)
  The scale consists of 32 items and comprises eight subscales. A higher score indicates higher levels of interoceptive awareness.
the Multidimensional Assessment of Interoceptive Awareness scale | six months after T2 (T3)
  The scale consists of 32 items and comprises eight subscales. A higher score indicates higher levels of interoceptive awareness.
the Multidimensional Assessment of Interoceptive Awareness scale | one year after T2 (T4)
  The scale consists of 32 items and comprises eight subscales. A higher score indicates higher levels of interoceptive awareness.
Wrist ActiGraph GT9X (ActiGraph, Pensacola, USA) | at baseline (T1)
  Participants will be asked to put on this ActiGraph GT9X (like a watch) on the wrist of the non-dominant hand for one week. Wrist ActiGraph GT9X is used to assess the average total sleep time (hours) per night.
Wrist ActiGraph GT9X (ActiGraph, Pensacola, USA) | In the 8th week from baseline (T2)
  Participants will be asked to put on this ActiGraph GT9X (like a watch) on the wrist of the non-dominant hand for one week. Wrist ActiGraph GT9X is used to assess the average total sleep time (hours) per night.
Wrist ActiGraph GT9X (ActiGraph, Pensacola, USA) | six months after T2 (T3)
  Participants will be asked to put on this ActiGraph GT9X (like a watch) on the wrist of the non-dominant hand for one week. Wrist ActiGraph GT9X is used to assess the average total sleep time (hours) per night.
Wrist ActiGraph GT9X (ActiGraph, Pensacola, USA) | one year after T2 (T4)
  Participants will be asked to put on this ActiGraph GT9X (like a watch) on the wrist of the non-dominant hand for one week. Wrist ActiGraph GT9X is used to assess the average total sleep time (hours) per night.

OTHER OUTCOMES:
the Chinese (Hong Kong) Short-Form-12 | at baseline (T1)
  A higher respective summary score indicates better levels of health.
the Chinese (Hong Kong) Short-Form-12 | In the 8th week from baseline (T2)
  A higher respective summary score indicates better levels of health.
the Chinese (Hong Kong) Short-Form-12 | six months after T2 (T3)
  A higher respective summary score indicates better levels of health.
the Chinese (Hong Kong) Short-Form-12 | one year after T2 (T4)
  A higher respective summary score indicates better levels of health.
the rumination subscale from the Rumination-Reflection Questionnaire | at baseline (T1)
  A higher score suggests greater ruminative tendencies.
the rumination subscale from the Rumination-Reflection Questionnaire | In the 8th week from baseline (T2)
  A higher score suggests greater ruminative tendencies.
the rumination subscale from the Rumination-Reflection Questionnaire | six months after T2 (T3)
  A higher score suggests greater ruminative tendencies.
the rumination subscale from the Rumination-Reflection Questionnaire | one year after T2 (T4)
  A higher score suggests greater ruminative tendencies.
the hyperarousal scale | at baseline (T1)
  A higher score suggests a higher arousal level.
the hyperarousal scale | In the 8th week from baseline (T2)
  A higher score suggests a higher arousal level.
the hyperarousal scale | six months after T2 (T3)
  A higher score suggests a higher arousal level.
the hyperarousal scale | one year after T2 (T4)
  A higher score suggests a higher arousal level.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan SH, Ng SM, Yu CH, Chan CM, Wang SM, Chan WC. The effects of an integrated mindfulness-based tai chi chuan programme on sleep disturbance among community-dwelling elderly people: protocol for a randomized controlled trial. Trials. 2022 Sep 24;23(1):808. doi: 10.1186/s13063-022-06737-4. PMID 36153623